CLINICAL TRIAL: NCT04024384
Title: Daratumumab as Maintenance After Peripheral Blood Stem Cell Transplantation From HLA-identical or Haploidentical Family Donor in the Treatment of Refractory or Relapsed Multiple Myeloma: a Phase 2 Trial
Acronym: DARALLO
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Promotor decision
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP180470
Record Dates: First submitted 2019-07-01; First posted 2019-07-18 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2019-07

CONDITIONS: Multiple Myeloma
Keywords: Myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daratumumab (Experimental): Daratumumab as maintenance after peripheral blood stem cell transplantation from HLA-identical or haploidentical family donor in the treatment of refractory or relapsed multiple myeloma
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — Daratumumab, 16 mg/kg, once a week for 8 weeks (cycles 1 and 2); then every 2 weeks for 16 weeks (cycles 3-6), then every 4 weeks thereafter (cycles 7-12).

SUMMARY:
The present protocol aims to test, whether an approach using (i) a reduced-toxicity TBF followed by a (ii) Daratumumab maintenance and (iii) prophylactic infusion of donor lymphocytes (pDLI), will be able to improve progression-free survival of patients with refractory or relapsed MM. This trial represents the first prospective protocol aiming to test the use of Daratumumab maintenance after HLA-identical or haploidentical allo-SCT in patients with MM.

DETAILED DESCRIPTION:
Allogeneic stem cell transplantation in patients with multiple myeloma (MM) Outcomes for patients with MM who are resistant to proteasome inhibitors (bortezomib) and immunomodulatory drugs (lenalidomide, thalidomide) are dramatically poor. The median expected overall survival (OS) in these patients is 9 months. New drugs such as pomalidomide or carfilzomib, when used in monotherapy, can only offer a median progression free survival (PFS) of 3.8 months and OS of 11.9 and 13.4 months, respectively.

Allogeneic stem cell transplantation (allo-SCT) remains the most reasonable treatment option, apart from palliative care, in patients with refractory or relapsed MM. No other strategy is able to offer any chance of cure for a patient at this stage. However, in the context of standard myeloablative (MAC) allo-SCT, results are limited in terms of feasibility in the larger patients' population who is in need, and by both a relatively high relapse incidence (RI) and especially high non-relapse mortality (NRM). Also, in the last decade, the advent of reduced intensity conditioning (RIC) allo-SCT and the improvement in supportive care management regarding infectious complications allowed a significant reduction of NRM. RIC expanded the transplant option to those patients who are ineligible for standard MAC allo-SCT either because of age or because of pre-existing comorbid conditions. While NRM is over 40% with MAC, relapse incidence remains high with either RIC or MAC. The major reason for treatment failure after allo-SCT for MM has become relapse, which is between 38% and 55%. Median PFS ranges from 10% to 32%. Thus, strategies to prevent relapse after allo-SCT for MM remain an unmet medical need.

Post-transplant maintenance therapy Consolidation/maintenance post-transplantation for MM has demonstrated to not only upgrade but also deepen the response, which translates into improved PFS. Studies investigated immunomodulatory drugs, thalidomide or lenalidomide, as maintenance therapy after allo-SCT. The observed activation of natural killer and regulatory T cells induced by immunomodulatory drugs provides an attractive rationale for its use post-transplant. But some concerns are raised by a high rate of graft-versus-host disease (GVHD) induction. In the prospective HOVON 76 trial, 43% patients stopped lenalidomide maintenance because of development of GVHD, 17% patients because of other adverse events, and 17% patients because of progression. Thus, lenalidomide maintenance after RIC allo-SCT in MM patients is not feasible, mainly because of the toxicity and the induction of acute GVHD.

Daratumumab, a human IgG1 monoclonal antibody that binds CD38-expressing malignant cells with high affinity and induces tumor cell death, has recently shown promising results in a phase 2 trial. Daratumumab was well tolerated, median PFS was 3.7 months and median duration of response was 7.4 months in patients who were refractory to both proteasome inhibitors and immunomodulatory drugs. Our first pilot experience, based on 3 patients with refractory MM suggests that Daratumumab maintenance is feasible. No grade 3-4 toxicities were observed. None of the patients experienced GVHD. After a median follow-up of 12 months, none of these patients relapsed. Thus, Daratumumab appears to be the ideal candidate to propose immunotherapy maintenance and reinforce the post-transplant immunomodulation strategy.

Prophylactic donor lymphocyte infusions Given that relapsed or refractory patients are at very high risk of relapse, prophylactic donor lymphocyte infusion (pDLI) is a promising approach to prevent relapse after allo-SCT. pDLI can improve remission status in 54% of the patients and result in 5-year PFS of 79%. The incidence and severity of acute GVHD remains manageable.

Type of donor Haploidentical family donors allow finding a quickly available donor for a majority of patients. T-cell replete haploidentical allo-SCT has now become feasible with the use of post-graft Cyclophosphamide, which reduces the risk of GVHD. In patients with relapsed or refractory hematologic malignancies, studies show no significant difference in terms of toxicity and outcomes between patients undergoing allo-SCT from a HLA-identical sibling and a haploidentical donor. Compared with unrelated donors, the outcomes are improved in haploidentical recipients. Thus, for these advanced patients, one should look first for a related donor, either matched or haploidentical. Searching for an unrelated donor may delay the procedure, with a risk of losing the opportunity for transplantation, and may be associated with worse outcomes compared with haploidentical allo-SCT.

Few studies have reported the outcomes of patients with MM after haploidentical allo-SCT. The most encouraging results have been reported with the RIC associating thiotepa, busulfan and fludarabine (TBF) in patients with heavily pretreated MM. The median 18-month PFS, OS and NRM were 33%, 63% and 10%, respectively.

The present protocol aims to test, whether an approach using (i) a reduced-toxicity TBF followed by a (ii) Daratumumab maintenance and (iii) prophylactic infusion of donor lymphocytes (pDLI), will be able to improve progression-free survival of patients with refractory or relapsed MM. This trial represents the first prospective protocol aiming to test the use of Daratumumab maintenance after HLA-identical or haploidentical allo-SCT in patients with MM.

This is a prospective, multicenter, open, non-randomized Phase II study that will include a total number of 38 patients included over a period of 2 years.

The population of the study is women and men adults (18-70 years) with refractory or relapsed multiple myeloma.

Treatment period will be 12 months Duration of inclusions will be 24 months So, total study duration (eg. 12 months after inclusion of last patient)will be 36 months

Each patient will receive: Daratumumab, 16 mg/kg, once a week for 8 weeks (cycles 1 and 2); then every 2 weeks for 16 weeks (cycles 3-6), then every 4 weeks thereafter (cycles 7-12).

A Patient is only eligible if:

* Absolute neutrophil count > 1 G/L
* Haemoglobin concentration > 7.5 g/dL
* Platelets > 50 G/L
* Estimated glomerular filtration rate > 20 mL/min according to CDK-EPI
* Is free of grade 2-4 acute GVHD since >30 days
* Is free of active infections

Is an interim analysis planned, if yes, list and specify timing(s): no Final study report timing after Last Patient, Last Visit: 3 months Publication submission timing after final study report: 3 months

The primary objective is to demonstrate that PFS at 12 months is higher than 40%. The trial would be designed to test the hypothesis P < 20% versus P>40% with one sided type I error rate 5% and power 80%. Using a one step A'Hern procedure, 35 patients should be transplanted. The analysis will be based on a binomial test comparing the observed 12 months PFS to 40%. In all, 38 patients will be included (taking into account that after registration, there is a risk of dropout i.e. patients, who will not receive a transplant due to rapidly progressive disease, infection or other events occurring after identification of a donor, but before start of conditioning).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of multiple myeloma
* Disease who progressed on salvage therapy or progressed within 60 days of the last treatment in patients who previously achieved at least a minimal response to treatment
* Stable disease or better 1 month before transplantation
* Age > 18 and < 70 years.
* Availability of an HLA-haploidentical or HLA-identical family donor
* Written informed consent.

Exclusion Criteria:

* Presence in the patient of donor HLA-specific antibodies (DSA) directed against the HLA haplo-identical family donor
* Karnofsky score <70%
* HIV positive patient, chronic or active Hepatitis B or Hepatitis C
* Life expectancy less than one month according to the attending physician
* Acute or chronic heart failure (Cardiac ejection fraction < 40%)
* Pulmonary function - diffusion capacity < 50% predicted
* Estimated glomerular filtration rate < 30 ml/min (CKD-EPI)
* Severe neurological or psychiatric disorders
* Any circumstances that preclude the use of the drugs used within the protocol
* Prior allogeneic stem cell transplantation
* Pregnancy or denied of effective contraceptive method

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
safety and efficacy of Daratumumab assessed by free survival | 1-year progression free survival in such patients
  The primary objective is to assess the 1-year progression free survival in such patients. If the smallest response proportion (pnew=0.4) could be achieved compare to the lowest response probability of interest (phypo=0.2), the treatment strategy would worth to be developed further.

SECONDARY OUTCOMES:
Disease response rate | day +30, day +90 and 12 months after transplantation
  Disease response rate at day +30, day +90 and 12 months after transplantation
Overall survival | 12 months after transplantation
  Overall survival, at 12 months after transplantation
GVHD-free | 12 months after transplantation
  GVHD-free, at 12 months after transplantation
Relapse-free survival | 12 months after transplantation
  Relapse-free survival at 12 months after transplantation
Cumulative incidence of relapse, death from disease, and non-relapse mortality | 12 months after transplantation.
  Cumulative incidence of relapse, death from disease, and non-relapse mortality within the first 12 months after transplantation.
Cumulative incidence of chronic GVHD as assessed by NIH Consensus Criteria | 12 months after transplantation.
  Cumulative incidence of chronic GVHD as assessed by NIH Consensus Criteria within the first 12 months after transplantation.
Serious adverse events of Daratumumab and number of infusion per patient | 12 months after transplantation.
  Serious adverse events of Daratumumab and number of infusion per patient
Serious adverse events of prophylactic donor lymphocytes infusion (pDLI) and number of infusion per patient | 12 months after transplantation.
  Serious adverse events of prophylactic donor lymphocytes infusion (pDLI) and number of infusion per patient
Quality of Life | at day-7, +30, +90, +180 and +360
  Quality of Life at day-7, +30, +90, +180 and +360
immune response analysis | (before transplant, 30 days after transplant, 1 year after transplant and in case of disease relapse)
  immune response analysis (before transplant, 30 days after transplant, 1 year after transplant and in case of disease relapse)

CONTACTS AND LOCATIONS:
Overall Officials: Rémy Dulery, PHD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service d'hématologie clinique et thérapie cellulaire, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided